CLINICAL TRIAL: NCT01597544
Title: Post-operative Voiding Dysfunction: the Preferred Method for Catheterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 241110
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2016-07

CONDITIONS: Voiding Dysfunction After Pelvic Organ Prolapse Surgery
Keywords: Voiding dysfunction; bladder catheter; prolapse surgery; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CISC instruction post-operatively (No Intervention): For those patients that are randomized to CISC instruction before surgery, instruction will begin on post-operative day one. One of the nurses from the hospital gynecology unit will teach and supervise the patients until they feel comfortable with the technique or until catheterization is no longer required (e.g. when the patient passes her voiding trial on two separate occasions). This is the protocol currently in use at our institution.
- CISC instruction pre-operatively (Active Comparator): Patients allocated to the pre-operative CISC teaching group will be taught how to perform CISC by one of urogynecology nurses working at the Women's Health Care Centre. Patients will be allowed to practice until they feel comfortable with the technique. This should take approximately 30 minutes. The session will take place on the day of their pre-operative medical appointment (PAF), which normally occurs less than a month before the surgery. If a patient is not seen in PAF or is seen more than a month before her surgery, a separate appointment for CISC teaching during the month preceding the surgery will be organized. Post-operatively, a nurse from the hospital gynecology unit will review the technique to make sure the patient is still comfortable with performing CISC.
  Interventions: Procedure: CISC instruction pre-operatively

INTERVENTIONS:
Procedure: CISC instruction pre-operatively — Patients allocated to the pre-operative CISC teaching group will be taught how to perform CISC by one of urogynecology nurses working at the Women's Health Care Centre. Patients will be allowed to practice until they feel comfortable with the technique. This should take approximately 30 minutes. The session will take place on the day of their pre-operative medical appointment (PAF), which normally occurs less than a month before the surgery. If a patient is not seen in PAF or is seen more than a month before her surgery, a separate appointment for CISC teaching during the month preceding the surgery will be organized. Post-operatively, a nurse from the hospital gynecology unit will review the technique to make sure the patient is still comfortable with performing CISC.
  Arms: CISC instruction pre-operatively

SUMMARY:
This study is divided into two parts. The first part is a prospective observational study of patients undergoing pelvic organ prolapse (POP) surgery. The goal is to determine patient preference between 3 different methods of bladder drainage in case of post-operative voiding dysfunction (POVD): transurethral indwelling catheterization (TIC), clean intermittent self-catheterization (CISC), and suprapubic tube (SPT). The second part of the study will be for those that choose CISC as their preferred method, whereby these patients will be randomized to receive CISC instruction either pre- or post-operatively to determine whether there is a difference in overall patient satisfaction based on timing of teaching.

The investigators hypothesize that patients that receive informed consent pre-operatively will favour the use of SPT over TIC and CISC to manage potential POVD.

Among those patients who opted for CISC in management of their post-operative voiding dysfunction, patients that are taught how to perform CISC pre-operatively in the clinic will have a higher level of satisfaction compared to those that are taught post-operatively in the hospital.

DETAILED DESCRIPTION:
Method PART 1 For the first part of the study, patient preference between TIC, CISC, SPT will be assessed during a face-to-face interview after the patient has had sufficient time to read the information sheet about the three options available and has had the opportunity to ask questions. This will ensure that every patient will receive the same information. The face-to-face interview will be performed by the patient's physician or by one of the two urogynecology nurses working at the St. Michael's Hospital Women's Health Care Centre. The patient's choice will be recorded in the pre-operative record and then in the study database by one of the study personnel.

Other data collected will include patient demographics (age, education level, level of home support, current or past occupation), clinical characteristics (BMI, parity, International Continence Society (ICS) stage of prolapse, and any pre-operative urinary diagnoses) (Appendix 4).

Peri-operatively, data collected will include the surgery performed, the length of hospital stay, and the occurrence of any peri-operative complications. At our institution we have defined normal voiding function as having a voided volume of > 200 mL with a post-voided residual (PVR) of < 100 mL or having a voided volume of > 400 mL with a PVR of < 33% (1/3) of the total voided volume. Patients have to meet these criteria on two separate voids while in hospital or they will be classified as having post-operative voiding dysfunction. Once they meet the criteria for voiding dysfunction, then the method of bladder drainage used (TIC, CISC and SPT) and the length of time it was used for will be recorded.

To reduce the rate of bacteriuria and other signs of bladder infection [25], antibiotic prophylaxis will be administered as usual to all patients that require bladder drainage for more than 24 hours. The antibiotic regimen consist of: Macrodantin 100 mg PO daily for the time of the bladder drainage, or Trimethoprim 100 mg PO daily if allergic. This is the regimen currently being used in our department.

For those patients that underwent catheterization in the post-operative period, satisfaction with regard to catheter management will be assessed using a visual analog scale based on a previously published questionnaire. This questionnaire will be administered on the day of discharge, on post-operative day seven, and six weeks after surgery. Post-operative bladder function in those that required catheterization will be assessed on post-operative day seven and six weeks after surgery using uroflowmetry testing, PVR measurement, and a specimen for urine culture.

PART 2 Women that were consented for the second part of the study will be randomized to either pre-operative CISC teaching in the clinic or post-operative CISC teaching in the hospital. A computer-generated list of random numbers will be used to allocate participants into 2 groups of equal size. To ensure consistency in teaching patients on CISC, nurses in the clinic and in the hospital will use the same protocol for instruction of CISC.

Patients allocated to the pre-operative CISC teaching group will be taught how to perform CISC by one of urogynecology nurses working at the Women's Health Care Centre. Patients will be allowed to practice until they feel comfortable with the technique. This should take approximately 30 minutes. The session will take place on the day of their pre-operative medical appointment (PAF), which normally occurs less than a month before the surgery. If a patient is not seen in PAF or is seen more than a month before her surgery, a separate appointment for CISC teaching during the month preceding the surgery will be organized. Post-operatively, a nurse from the hospital gynecology unit will review the technique to make sure the patient is still comfortable with performing CISC.

Patients allocated to the post-operative CISC teaching group will be instructed on CISC after surgery, starting on post-operative day one. One of the nurses from the hospital gynecology unit will teach and supervise the patients until they feel comfortable with the technique or until catheterization is no longer required (e.g. when the patient passes her voiding trial on two separate occasions). This is the protocol currently in use at our institution.

Patients in both groups will have to be comfortable and independent in performing CISC prior to being discharged from the hospital. Following their discharge, a nurse from the Women's Health Care Centre will be available to answer any questions by telephone.

For both groups, satisfaction will be assessed with a questionnaire that will be administered on the day of discharge, on post-operative day seven, and six weeks after surgery. Assessment of post-operative bladder function in those that required catheterization will occur on post-operative day seven and six weeks after surgery using uroflowmetry testing, PVR measurement, and a specimen for urine culture.

Patients with no post-operative voiding dysfunction will be withdrawn from the study. Since it is impossible to predict who will experience post-operative voiding dysfunction, it is essential to recruit all potential participants prior to surgery so that they can receive pre-operative CISC teaching if allocated to this group. Pre-operative data, however, will be kept for all recruited patients for the purose of study analyses.

Data analysis PART 1 Demographic measures, catheterization choice, and clinical data will be summarized using descriptive statistics. Patient satisfaction will be assessed using questionnaires that will be reviewed and scored. The questionnaire has 6 items and each item consist of a 10 cm line visual analogue scale. Patients will be asked to put an "X" on this line between the 2 extremes. The distance from the beginning of the line to the patient's X will be measured and the score will be obtained. Scores will be calculated by adding the scores of the 6 items (range 0 to 60), then dividing by 6 and multiplying by 10. Missing items are dealt with by using the sum from answered items only, dividing by the number of items answered. Patient who answered fewer than 4 questions will not be considered in the analyses.

PART 2 As above, demographic measures and clinical data will be summarized using descriptive statistics. Each of the questionnaires will be reviewed and scored. For this part of the study, the questionnaire has been modified with the addition of three items with a response scale score of 0 to 10. Scores are calculated by adding the scores of the 9 items (range 0 to 90), then dividing by 9 and multiplying by 10. Missing items are dealt with by using the Sum from answered items only, dividing by the number of items answered. Patient who answered fewer than 6 questions will not be considered in the analyses. Each of the questionnaires will be reviewed and scored. Satisfaction scores between the two groups (pre-operative and post-operative teaching) will be compared using a two-sided Student's t-test.

For both parts of the study, continuous variables will be summarized as means (standard deviation) or medians (minimum, maximum) and compared between groups using Student's t-tests or Kruskal Wallis tests. Categorical variables will be summarized as counts (percent) and compared between groups using Fisher's exact tests.

Sample Size Calculation For the first part of the study, we are aiming to survey a minimum of 150 patients. The power calculation for the second part of the study is based on a previous study [11]. Based on these findings, we defined the minimal relevant difference in patient satisfaction with regard to CISC teaching to be 30% with a standard deviation of +/- 30. With a power of 0.8 and an alpha of 0.05, the minimum number of patients required in each group is eight. We anticipate a 10% drop out rate after consent and we expect that 65% of patients will not require any form of outpatient catheterization after their surgery. Therefore, we will require 25 patients per arm for the second part of the study. Recruitment for the first part of the study will cease once we have recruited all the patients required for the second part or once we have recruited 150 patients, whichever comes first.

Timeline for completion Based on the operative hospital data from 2010, we will need approximately 24 months to recruit patients and collect data. Three more months will be required for data analysis and manuscript preparation.

ELIGIBILITY:
Inclusion Criteria:

* All pre-operative patients seen at the St. Michael's Hospital Women's Health Care Centre and consented for a POP surgery will be eligible to participate in the first part of this study.
* All patients undergoing POP surgery that choose CISC as their preferred method of bladder drainage will then be eligible for the second part of the study.
* Additional inclusion criteria for both parts of the study include: female gender, greater than 18 years of age, and able to read and write in the English language

Exclusion Criteria:

* Significant cognitive impairment, a history of neurogenic voiding dysfunction, a history of prior catheter use in the outpatient setting, as well as any patients undergoing outpatient surgery or surgery that only includes the posterior vaginal compartment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Part 1: Patient catheter preference | 24 months
  For the first part of the study, the primary outcome is determining patient preference for method of bladder drainage for potential post-operative voiding dysfunction when asked pre-operatively. They will be given the options of either transurethral indwelling catheter (TIC), clean intermittent self catheterization (CISC), or suprapubic tube (SPT).
Part 2: patient satisfaction with regard to timing of CISC teaching. | 24 months
  For the second part of the study, the primary outcome measure is the difference in patient satisfaction levels between those that had pre-operative CISC teaching compared with those that had the standard post-operative CISC teaching.

SECONDARY OUTCOMES:
Patient satisfaction with catheter choice | 24 months
  This will be assessed using a visual analog scale based on a previously published questionnaire. This questionnaire will be administered on the day of discharge, on post-operative day seven, and six weeks after surgery. This will be compared between the three different catheter groups.
Incidence of post-operative voiding dysfunction after prolapse surgery | 24 months
  We will determine the actual number of patients that required catheter use to manage acute voiding dysfunction after prolapse surgery.
Bladder function after catheter use | 24 months
  We will assess bladder function in those patients that required bladder catheterization to manage post-operative voiding dysfunction by performing uroflowmetry and post-void residual measurements at one and six weeks after surgery. This will be compared between the three different catheter groups.
Incidence of bacteruria/urinary tract infection after catheter use | 24 months
  We will assess the incidence of bacteruria/urinary tract infection in those patients that required bladder catheterization to manage post-operative voiding dysfunction by performing uroflowmetry and post-void residual measurements at one and six weeks after surgery. This will be compared between the different catheter groups.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen D McDermott, MD, FRCSC, Principal Investigator — St. Michael's Hospital, University of Toronto
Locations (1):
- St. Michael's Hospital, University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hakvoort RA, Dijkgraaf MG, Burger MP, Emanuel MH, Roovers JP. Predicting short-term urinary retention after vaginal prolapse surgery. Neurourol Urodyn. 2009;28(3):225-8. doi: 10.1002/nau.20636. PMID 19130599
- [Background] Schiotz HA. Comparison of 1 and 3 days' transurethral Foley catheterization after retropubic incontinence surgery. Int Urogynecol J Pelvic Floor Dysfunct. 1996;7(2):98-101. doi: 10.1007/BF01902381. PMID 8798095
- [Background] Glavind K, Morup L, Madsen H, Glavind J. A prospective, randomised, controlled trial comparing 3 hour and 24 hour postoperative removal of bladder catheter and vaginal pack following vaginal prolapse surgery. Acta Obstet Gynecol Scand. 2007;86(9):1122-5. doi: 10.1080/00016340701505317. PMID 17712655
- [Background] Hakvoort RA, Elberink R, Vollebregt A, Ploeg T, Emanuel MH. How long should urinary bladder catheterisation be continued after vaginal prolapse surgery? A randomised controlled trial comparing short term versus long term catheterisation after vaginal prolapse surgery. BJOG. 2004 Aug;111(8):828-30. doi: 10.1111/j.1471-0528.2004.00181.x. PMID 15270931
- [Background] Van Der Steen A, Detollenaere R, Den Boon J, Van Eijndhoven H. One-day versus 3-day suprapubic catheterization after vaginal prolapse surgery: a prospective randomized trial. Int Urogynecol J. 2011 May;22(5):563-7. doi: 10.1007/s00192-011-1358-7. Epub 2011 Mar 3. PMID 21369817
- [Background] Alonzo-Sosa JE, Flores-Contreras JT, Paredes-Canul M. [Method for transurethral catheterization for 1-3 days for pelvic floor relaxation in the postoperative period]. Ginecol Obstet Mex. 1997 Nov;65:455-7. Spanish. PMID 9441144
- [Background] Guzman S, Israel E, Puente R, Iglesias R, Rosa G, Ulloa C. [Handling of Foley catheter regarding urinary retention syndrome following vaginal surgery]. Rev Chil Obstet Ginecol. 1994;59(4):280-3. Spanish. PMID 7659824
- [Background] Bidmead J, Cardozo L. Retropubic urethropexy (Burch colposuspension). Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(4):262-5. doi: 10.1007/s001920170050. PMID 11569656
- [Background] Colombo M, Vitobello D, Proietti F, Milani R. Randomised comparison of Burch colposuspension versus anterior colporrhaphy in women with stress urinary incontinence and anterior vaginal wall prolapse. BJOG. 2000 Apr;107(4):544-51. doi: 10.1111/j.1471-0528.2000.tb13276.x. PMID 10759276
- [Background] Kleeman S, Goldwasser S, Vassallo B, Karram M. Predicting postoperative voiding efficiency after operation for incontinence and prolapse. Am J Obstet Gynecol. 2002 Jul;187(1):49-52. doi: 10.1067/mob.2002.124841. PMID 12114887
- [Background] Jannelli ML, Wu JM, Plunkett LW, Williams KS, Visco AG. A randomized controlled trial of clean intermittent self-catheterization versus suprapubic catheterization after urogynecologic surgery. Am J Obstet Gynecol. 2007 Jul;197(1):72.e1-4. doi: 10.1016/j.ajog.2007.02.043. PMID 17618764
- [Background] Vierhout ME. Prolonged catheterization after vaginal prolapse surgery. Acta Obstet Gynecol Scand. 1998 Nov;77(10):997-9. PMID 9849844
- [Background] Kringel U, Reimer T, Tomczak S, Green S, Kundt G, Gerber B. Postoperative infections due to bladder catheters after anterior colporrhaphy: a prospective, randomized three-arm study. Int Urogynecol J. 2010 Dec;21(12):1499-504. doi: 10.1007/s00192-010-1221-2. Epub 2010 Aug 4. PMID 20683580
- [Background] Dobbs SP, Jackson SR, Wilson AM, Maplethorpe RP, Hammond RH. A prospective, randomized trial comparing continuous bladder drainage with catheterization at abdominal hysterectomy. Br J Urol. 1997 Oct;80(4):554-6. doi: 10.1046/j.1464-410x.1997.t01-1-00376.x. PMID 9352691
- [Background] Woodward S, Rew M. Patients' quality of life and clean intermittent self-catheterization. Br J Nurs. 2003 Oct 9-22;12(18):1066-74. doi: 10.12968/bjon.2003.12.18.11782. PMID 14581839
- [Background] Maynard FM, Diokno AC. Urinary infection and complications during clean intermittent catheterization following spinal cord injury. J Urol. 1984 Nov;132(5):943-6. doi: 10.1016/s0022-5347(17)49959-9. PMID 6333518
- [Background] Kessler TM, Ryu G, Burkhard FC. Clean intermittent self-catheterization: a burden for the patient? Neurourol Urodyn. 2009;28(1):18-21. doi: 10.1002/nau.20610. PMID 18726939
- [Background] Hakvoort RA, Thijs SD, Bouwmeester FW, Broekman AM, Ruhe IM, Vernooij MM, Burger MP, Emanuel MH, Roovers JP. Comparing clean intermittent catheterisation and transurethral indwelling catheterisation for incomplete voiding after vaginal prolapse surgery: a multicentre randomised trial. BJOG. 2011 Aug;118(9):1055-60. doi: 10.1111/j.1471-0528.2011.02935.x. Epub 2011 Apr 11. PMID 21481147
- [Background] Scott BM. Clinical and cost effectiveness of urethral catheterisation: a review. J Perioper Pract. 2010 Jul;20(7):235-40. doi: 10.1177/175045891002000701. PMID 20701200
- [Background] Niel-Weise BS, van den Broek PJ. Urinary catheter policies for short-term bladder drainage in adults. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD004203. doi: 10.1002/14651858.CD004203.pub2. PMID 16034924
- [Background] McPhail MJ, Abu-Hilal M, Johnson CD. A meta-analysis comparing suprapubic and transurethral catheterization for bladder drainage after abdominal surgery. Br J Surg. 2006 Sep;93(9):1038-44. doi: 10.1002/bjs.5424. PMID 16804872
- [Background] Park HC, Son JH, Jang SH. Rethinking suprapubic cystostomy in voiding dysfunction: new trial with timed drainage. Korean J Urol. 2010 Dec;51(12):847-52. doi: 10.4111/kju.2010.51.12.847. Epub 2010 Dec 21. PMID 21221205
- [Background] Dunn TS, Figge J, Wolf D. A comparison of outcomes of transurethral versus suprapubic catheterization after Burch cystourethropexy. Int Urogynecol J Pelvic Floor Dysfunct. 2005 Jan-Feb;16(1):60-2; discussion 62. doi: 10.1007/s00192-004-1209-x. Epub 2004 Jul 28. PMID 15647964
- [Background] Stekkinger E, van der Linden PJ. A comparison of suprapubic and transurethral catheterization on postoperative urinary retention after vaginal prolapse repair: a randomized controlled trial. Gynecol Obstet Invest. 2011;72(2):109-16. doi: 10.1159/000323827. Epub 2011 Feb 18. PMID 21335940
- [Background] Niel-Weise BS, van den Broek PJ. Antibiotic policies for short-term catheter bladder drainage in adults. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD005428. doi: 10.1002/14651858.CD005428. PMID 16034973